CLINICAL TRIAL: NCT05712616
Title: Role of Strontium Ranelate in Radiological Healing of Proximal Femur Fractures. A Phase IV Double Blinded Randomized Controlled Trial
Brief Title: Role of Strontium Ranelate in Proximal Femur Fragility Fractures.
Acronym: STRONG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Collaborators: AO Trauma Middle East and North Africa (Unknown)
Responsible Party: Principal Investigator, Dr. Marij Zahid, Instructor orthopedic surgery, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6189
Record Dates: First submitted 2022-10-28; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Fragility Fracture; Femur; Fracture, Pertrochanteric; Clinical Trial
MeSH Terms: conditions — Fractures, Bone | interventions — strontium ranelate; lacto-N-hexaose; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strontium group (Active Comparator): Trial drug given in the form of sachet 2gm/sachet once every day
  Interventions: Drug: Strontium Ranelate
- Placebo (Lactose) (Placebo Comparator): Look, smell, taste alike lactose 2gm/sachet in form of sachet
  Interventions: Drug: Lacto-N-Hexaose

INTERVENTIONS:
Drug: Strontium Ranelate — Dual mode of action, anabolic and anti-resorptive
  Other Names: placebo
  Arms: Strontium group
Drug: Lacto-N-Hexaose — Placebo look alike drug
  Other Names: Lactose
  Arms: Placebo (Lactose)

SUMMARY:
This study is being conducted with the aim of comparing the time to bone healing after surgery for fragility fractures of proximal femur between patients receiving strontium ranelate and placebo. Patients recruited are of 60 years of age and above. Bone healing will be assessed on clinical parameters when patient is able to ambulate full weight bearing without pain and on Xray images using RUSH score. Moreover Dexa scan will be performed pre-operatively and at 3 months postoperatively. The findings of this study will help in setting up guidelines for treatment of fragility proximal femur fractures in our population as there is still paucity of literature on effectiveness of strontium ranelate from our part of the world.

ELIGIBILITY:
Inclusion Criteria:

* All patients with age =/> 60 years with proximal femur fracture including per-trochanteric, sub-trochanteric and neck of femur fractures amnebale to ORIF.
* ORIF will include hip cannulated screws, dynamic hip screw and intra-medullary nails.

Exclusion Criteria:

* Patients with metabolic bone diseases.
* Patients with pathological fractures like tumor, osteopetrosis etc.
* Patients with prior Ischemic heart diseases and underwent PCI or CABG

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
change in Radiological healing on radiographs | 12 weeks and 24 weeks
  Difference in RUSH (Radiological Healing score for hip) score measured at 12 weeks and 24 weeks

SECONDARY OUTCOMES:
change Bone mineral density through DEXA scan | pre-operatively or peri-admission and at 3 months
  Difference in bone density T scores between pre-op and 3 months studies

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided